CLINICAL TRIAL: NCT03950284
Title: Assessment of the Stability of Immediately Loaded Dental Implants With the All-on-four Technique in Free Vascularized Fibular Grafts Used for Reconstruction of the Jaws
Brief Title: Assessment of the Stability of Immediately Loaded All-on-four Dental Implants in FFF Used for Reconstruction of the Jaws
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Shawky, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cairo omfs masters
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Reconstructed Jaws; Free Fibula Flaps; All on Four Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immediate loading with all on four technique in FFF (Experimental): immediately loaded dental implants with the all-on-four technique in free vascularized fibular grafts
  Interventions: Device: immediate loading with all on four technique in FFF

INTERVENTIONS:
Device: immediate loading with all on four technique in FFF — All cases will undergo surgery under local regional anesthesia. Injection of local anaesthesia (Articaine 4% and 1:100000 epinephrine) for regional infiltration. Sequential drilling then insertion of the dental implant fixtures and abutments on which the prefabricated temporary prosthesis will be fixed.

SUMMARY:
The use of free vascularized fibula flaps for bony reconstruction has proved its success as a substitution for the resected bone and in some instances, the surrounding soft tissues

The aim of this case series study is to evaluate the stability of the dental implants placed in free fibula flaps substituting a resected mandible and/or maxilla when they are immediately loaded with the All-On-Four technique along with the patient satisfaction.

DETAILED DESCRIPTION:
• Preoperative phase :

Patients will be subjected to:

* Case history including personal data, medical, surgical and family history.
* Clinical examination
* Radiographic examination using computed tomography (C.T) bony and soft tissue window.
* Diagnostic studying casts.
* Operative phase :

All cases will undergo surgery under local regional anesthesia. Injection of local anaesthesia (Articaine 4% and 1:100000 epinephrine) for regional infiltration. Sequential drilling then insertion of the dental implant fixtures and abutments on which the prefabricated temporary prosthesis will be fixed.

• Postoperative care Proper postoperative instructions will be given to the patient such as strict oral hygiene measures and soft diet for 1 month, in addition to the postoperative medications including antibiotics (amoxicillin 1g capsules b.d.s ) and analgesics (diclofenac potassium 50mg as needed). Adherence to follow ups will be also instructed

ELIGIBILITY:
Inclusion Criteria

* Patients with reconstructed jaws with free fibula flaps in either or both jaws.
* Age group : from 15 to 60 years old
* No sex predilection
* Patients with no contraindications to surgical intervention Exclusion Criteria
* Patients with systemic condition counteracting with the surgical procedure.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Primary Stability | 6 months
  The primary outcome is the implant stability determined by the insertion torque at the time of insertion using OSSTELL device

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shawky, MSc, Principal Investigator — Assistant lecturer. OMFS. Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt